CLINICAL TRIAL: NCT04955314
Title: The Importance of Manual Therapy Specificity Referred to Pain Intensity in Patients With Subacute and Unspecified Low Back Pain
Brief Title: Value of Manual Therapy Specificity Referred to Pain Intensity in Patients With Subacute and Unspecified Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Physiotherapist, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2020/6/56
Record Dates: First submitted 2021-06-02; First posted 2021-07-08 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Low Back Pain
Keywords: low back pain; subacute; manual therapy; PA; mobilization; manipulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The patients will be divided into two groups and a different physiotherapist from the one who will subsequently perform the intervention will assess and determine which is the most painful segment in each of them.
  In the first of the groups, the intervention to be carried out will be through posteroanterior vertebral mobilizations in the most painful lumbar segment. The members of the second group will undergo this same technique on a painful segment of the region adjacent to the one they have referred as the main source of pain.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PA mobilizations on their main painfull vertebral segment (Experimental): Patients who will be treated with PA mobilizations on their main painfull vertebral segment.
  Interventions: Other: PA vertebral mobilization
- PA mobilizations on an adjacent vertebral segment from the most painful (Experimental): Patients who will be treated with PA mobilizations on an adjacent vertebral segment from the most painful.
  Interventions: Other: PA vertebral mobilization

INTERVENTIONS:
Other: PA vertebral mobilization — A PA mobilization is a technique in which one vertebra slides over another due to a force applied with the hands of the physiotherapist

SUMMARY:
This study proves the specificity of manual therapy in unspecified an subacute low back pain

DETAILED DESCRIPTION:
The purpose of the study is to determine the importance of manual therapy specificity in relation to subacute low back pain.

In order to do this, it will be selected a sample of at least 48 people who suffer low back pain whose duration has not exceeded 12 weeks. Patients will be divided into two groups and a different physiotherapist from the one who will subsequently perform the intervention, will assess and determine which is the most painful segment in each of them.

In the first group, the intervention to be carried out will be through posteroanterior (PA) vertebral mobilizations in the most painful lumbar segment. The members of the second group will undergo this same technique on a painful segment of the region adjacent to the one they have referred as the main source of pain.

Each of these sessions will continue until the patient's symptoms have decreased two points on the numerical scale of pain. There will be one session per week, for six weeks.

To determine the differences between the two groups, there will be carried out 4 measurements of pain, functional disability, quality of life and kinesiophobia, and 3 measurements of pressure pain threshold were performed. Each one of them will be carried out in the first session, in the third week of treatment, in the last session of the treatment and one month after the end of the treatment. The last measeurement will be executed online and that is why the pressure pain threshold will be measured three times while the rest will be do it.

The hypothesis is that it won´t be differences in the amount of pain between the tratment on the main painful segment and the treatment on his adyacent segment.

ELIGIBILITY:
Inclusion Criteria:

* People aged between 18 and 65 years old with unspecific and subacute low back pain.
* Participants must be capable of walking twice a week 20 minutes per day.

Exclusion Criteria:

* People with history of spinal surgeries, osteoporosis and tumor.
* Pregnant and people with severe respiratory and cardiac illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity | Baseline, 3 weeks, 6 weeks and 10 weeks after intervention beginning.
  Using Numeric Pain Rating Scale (NPRS). In this scale patients rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)

SECONDARY OUTCOMES:
Change in Health related quality of life | Baseline, 3 weeks, 6 weeks and 10 weeks after intervention beginning.
  Using SF-36.This scale is made up of 36 items divided into 8 sections. The result can range from 0 to 100, where 0 is the worst possible health condition and 100 is the best one.
Change in Kinesiophobia | Baseline, 3 weeks, 6 weeks and 10 weeks after intervention beginning.
  Using the tampa scale for kinesiophobia-11 (TSK-11) to measure fear of movement, pain and injury relapse. The result can range from 11-44 points where higher scores indicate greater fear of pain, movement, and injury.
Change in Disability | Baseline, 3 weeks, 6 weeks and 10 weeks after intervention beginning.
  Using Oswestry Disability Index (ODI).The final score of this scale ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound
Change in Pressure Pain Threshold | Baseline, 3 weeks and 6 weeks after intervention beginning.
  Using an Algometer. This is an instrument for measuring sensitivity to pressure or to pain

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Achalandabaso, Study Director — University of Jaen
Locations (1):
- Universidad de Alcalá, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No